CLINICAL TRIAL: NCT00742079
Title: Pilot Study of Pretreatment D-cycloserine for CBT-assessment of Paranoid Delusions in Schizophrenia
Brief Title: Using D-cycloserine to Enhance the Benefits of Cognitive Behavioral Therapy for Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50MH060450 (NIH); 2P50MH060450-07A1 (NIH); DATR A3-NSC (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Paranoid Schizophrenia; Paranoid Delusions; CBT; D-Cycloserine
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid | interventions — Cycloserine; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 D-cycloserine, placebo (Experimental): Participants will receive D-cycloserine 1 hour before a cognitive behavioral therapy (CBT) session on Week 1, and they will receive placebo 1 hour before a CBT session on Week 2.
  Interventions: Drug: D-cycloserine; Behavioral: Cognitive Behavioral Therapy
- 2 Placebo, D-cycloserine (Experimental): Participants will receive placebo 1 hour before a CBT session on Week 1, and they will receive D-cycloserine 1 hour before a CBT session on Week 2.
  Interventions: Drug: D-cycloserine; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: D-cycloserine — Single, fixed 50-mg dose of D-cycloserine administered 1 hour prior to a CBT session
  Other Names: Seromycin
Behavioral: Cognitive Behavioral Therapy — One-hour talk therapy session with a trained clinician aimed at increasing cognitive flexibility by examining alternative explanations to everyday situations
  Other Names: CBT

SUMMARY:
This study will examine whether pretreatment with D-cycloserine before cognitive behavioral therapy can reduce impairments still present in people with stable cases of schizophrenia as well as determine which traits make schizophrenics most likely to respond to D-cycloserine treatment.

DETAILED DESCRIPTION:
Schizophrenia is a debilitating chronic condition that affects approximately 1 % of Americans, who experience symptoms such as hallucinations, delusions, and disorders of thought and movement. These symptoms are described as positive symptoms, because they are experienced in addition to what healthy individuals experience. Negative symptoms, which are reductions in normal functioning, and cognitive deficits, which are problems in thinking, also plague people with schizophrenia. The negative symptoms and cognitive deficits associated with schizophrenia are produced in otherwise healthy people by neurotransmitters inhibiting the glutamatergic N-methyl-d-aspartate NMDA receptors in the brain. This inhibition of NMDA receptors also causes intensification of psychotic symptoms in otherwise stabilized schizophrenic patients. The drug D-cycloserine partially excites NMDA receptors, and it has been used to help patients with anxiety disorders to overcome phobias while they are receiving cognitive behavioral therapy. This study will examine whether D-cycloserine can increase the cognitive flexibility of someone undergoing CBT and thereby enhance the therapy's ability to reduce a patient's belief in paranoid delusions, preoccupation with delusions, and related distress.

All participants will be screened to ensure proper diagnosis of schizophrenia without other conditions. Those who pass will be randomly assigned to receive either D-cycloserine first or a placebo pill first. One week after the screening, participants in the D-cycloserine group will be given the drug before a 1-hour session of simulated CBT treatment. Those in the placebo condition will receive a placebo pill before an identical session. Two weeks after the screening, both groups will be called back for another session of CBT, but the pills they receive will be switched. Those who received D-cycloserine the first week will receive placebo, and those who received placebo will receive D-cycloserine. The CBT sessions will attempt to increase cognitive flexibility in patients by asking them to provide alternate explanations for common situations. At screening, at the start of visits on the first and second weeks, and at a follow-up visit on the third week, participants will undergo a series of assessments, including interviews, computerized tests, and self-report measures. Belief in, preoccupation with, and distress caused by delusions, as well as degree of cognitive flexibility, will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, schizoaffective disorder, or schizophrenia, paranoid subtype, based on chart review, Structured Clinical Interview for DSM-IV, and consultation with the patient's clinicians
* Medicated with an antipsychotic agent other than clozapine at a stable dose for at least 6 weeks
* Scores at least 3, or "moderate," on the Scale for the Assessment of Positive Symptoms global delusion rating
* Paranoid or referential delusional content
* Never engaged in formal CBT psychotherapy in the past

Exclusion Criteria:

* Diagnosis of a comorbid Axis I disorder other than schizophrenia
* Active substance abuse or dependence within 6 months
* Significant suicidal ideation within 6 weeks
* Pregnant or nursing
* Unstable medical disorder
* impaired renal clearance (creatinine <60mg/dL/min)
* Suffering from dementia
* Suffering from seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C. Goff, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Schizophrenia Program - Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gottlieb JD, Cather C, Shanahan M, Creedon T, Macklin EA, Goff DC. D-cycloserine facilitation of cognitive behavioral therapy for delusions in schizophrenia. Schizophr Res. 2011 Sep;131(1-3):69-74. doi: 10.1016/j.schres.2011.05.029. Epub 2011 Jun 30. PMID 21723096

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from an urban community mental health center in Boston, MA from September 2006 to May 2010.
Pre-assignment Details: 31 participants were screened, 10 were excluded (7 did not meet inclusion criteria and 2 refused to participate, 1 excluded for reasons not listed in study publication)
Groups:
- 1 D-cycloserine First, Then Placebo: Participants received 50 mg D-cycloserine 1 hour before a cognitive behavioral therapy (CBT) session on Week 1, and then received placebo 1 hour before a CBT session on Week 2.
- 2 Placebo First, Then D-cycloserine: Participants received placebo 1 hour before a CBT session on Week 1, and then received 50 mg D-cycloserine 1 hour before a CBT session on Week 2.
Period: Overall Study
Arm/Group | 1 D-cycloserine First, Then Placebo | 2 Placebo First, Then D-cycloserine
Started | 11 | 10
Baseline/Week 1 (Received Dose 1) | 11 | 9
Week 2 (Received Dose 2) | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 D-cycloserine, Then Placebo: Participants received 50 mg D-cycloserine 1 hour before a cognitive behavioral therapy (CBT) session on Week 1, and then received placebo 1 hour before a CBT session on Week 2.
- 2 Placebo, Then D-cycloserine: Participants received placebo 1 hour before a CBT session on Week 1, and then received 50 mg D-cycloserine 1 hour before a CBT session on Week 2.
- Total: Total of all reporting groups
Arm/Group | 1 D-cycloserine, Then Placebo | 2 Placebo, Then D-cycloserine | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (9.0) | 51.4 (13.0) | 50.2 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Alternative Beliefs Assessment
Description: Number of alternative beliefs generated on the Alternative Beliefs Assessment. This assessment used nine vignettes describing social interactions: three of neutral content, three negatively-valanced, and three tailored to the patient's specific delusions. Participants were asked to generate as many explanations (alternative beliefs) as they could for each scenario, and the number of explanations produced in response to each item was recorded. Scores could range from 0 to as many explanations a person could produce (no maximum value). The total score was calculated by adding all alternative beliefs generated from each vignette. A higher number of alternative beliefs generated reflects a greater degree of cognitive flexibility.
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- D-cycloserine: Participants receive 50 mg of D-cycloserine
- Placebo: Participants receive 50 mg of placebo
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 14.05 (12.71) | 10.70 (16.08)

2. Secondary Outcome: Change in Psychotic Rating Scales (PSYRATS) Delusion Score
Description: The Delusions subscale is a 6 item clinician administered scale, with Likert items 0-4 and range is 0-24. Higher scores represent worse outcomes
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale | -0.89 (2.49) | -0.47 (3.08)

3. Secondary Outcome: Change in Beck Cognitive Insight Scale (BCIS)
Description: The BCIS is a 15-item self-report scale with Likert items 0-3. It consists of a composite score, where higher scores represent better outcomes, and there are 2 subscales: 1) Self-Reflectiveness (higher scores represent better outcomes) and 2) Self-Certainty (higher scores represent worse outcomes). The total score for each scale is the sum of the item scores that comprise it (see below). The BCIS composite index is calculated as self-reflectiveness minus self-certainty.
  Step 1. Score every item on the BCIS from "0" to "3" according to the following rule:
  "Do Not Agree at All" = 0, "Agree Slightly" = 1, "Agree a Lot" = 2, "Agree Completely" = 3 Step 2. Calculate self-reflectiveness subscale: sum items 1, 3, 4, 5, 6, 8, 12, 14, and 15.
  Step 3. Calculate self-certainty subscale: sum items 2, 7, 9, 10, 11, and 13. Step 4. Calculate BCIS composite index: self-reflectiveness minus self-certainty.
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale
  Composite Score | -0.26 (3.46) | 0.44 (4.16)
  Self-Certainty Score | 0.11 (3.68) | -0.56 (2.64)
  Self-Reflectiveness Score | -0.16 (2.81) | -0.11 (3.23)

4. Secondary Outcome: Change in Bead Task Score Measuring Probabilistic Reasoning
Description: The Bead task is a reasoning task, where the number of beads guessed is the numeric value represented in the data. The lower end range is 1, and there is no upper range limit. Higher scores represent better outcomes.
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale | 0.45 (4.47) | 0.10 (5.16)

5. Secondary Outcome: Change in the Maudsley Assessment of Delusions Scale
Description: This scale is a one-question item added on to the Bead Task. The one item asks for a certainty rating, from 1-3. Higher scores represent better outcomes.
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale | 0.05 (0.40) | -0.16 (0.37)

ADVERSE EVENTS:
Time Frame: Three week period from baseline until week 2 of treatment.
Description: No adverse events were reported following ingestion of study drug.
Arm/Group | 1 D-cycloserine, Then Placebo | 2 Placebo, Then D-cycloserine
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
The cross-over design of this study produced results that are difficult to interpret due to a significant order effect. Larger and longer trials are needed to assess whether this treatment may benefit patients with medication resistant delusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No